CLINICAL TRIAL: NCT02960503
Title: Macrolide Therapy to Improve Forced Expiratory Volume in 1 Second in Adults With Sickle Cell Disease: a Feasibility Trial
Brief Title: Macrolide Therapy to Improve Forced Expiratory Volume in 1 Second in Adults With Sickle Cell Disease
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Key personnel moved to new location. Therefore, we had insufficient resources to initiate the trial.
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Michael DeBaun, Professor of Pediatrics and Medicine, Vice Chair for Clinical and Translational Research, J.C. Peterson Chair in Pediatric Pulmonology, Director, Vanderbilt-Meharry Center for Excellence in Sickle Cell Disease, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 161332
Record Dates: First submitted 2016-11-02; First posted 2016-11-09 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; pulmonary complications; reduced FEV1; azithromycin; lung function
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment arm (azithromycin) (Active Comparator): Treatment arm: azithromycin 500 mg three times a week for 6 months
  Interventions: Drug: Azithromycin
- Placebo arm (Placebo Comparator): Control arm: placebo three times a week for 6 months
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Azithromycin — Study participants will be randomized to the treatment arm (azithromycin 500 mg three times a week for 6 months).
  Other Names: Zithromax, zmax, z-pack
  Arms: Treatment arm (azithromycin)
Other: Placebo — Study participants will be randomized to the control arm (placebo three times a week for 6 months).
  Arms: Placebo arm

SUMMARY:
Sickle cell anemia (SCA) is a life-threatening, monogenic disorder associated with early death when compared to individuals without SCA. Pulmonary complications, namely acute chest syndrome, obstructive lung disease and pulmonary hypertension, are the most common causes of death in patients with SCA. Recent studies suggest that lung specific inflammation is a hallmark of SCA and underlies pulmonary pathology. To date, no therapy has been shown to improve the pulmonary complications of SCA. Macrolides have pleomorphic effects in the lung with improvement in pulmonary function, symptoms and inflammatory markers demonstrated in several inflammatory pulmonary conditions such as cystic fibrosis, asthma, COPD and post-transplant bronchiolitis obliterans. Investigators hypothesize that low dose macrolide therapy is well tolerated and can improve pulmonary function and symptoms in patients with SCA. The objective of this project is to assess the feasibility of macrolides to attenuate or reverse the decrease in %predicted FEV1 in adults with SCA in a single-site, randomized, placebo-controlled feasibility trial.

DETAILED DESCRIPTION:
Specific aim 1: To determine acceptability of a clinical trial in which participants are randomly allocated to either a placebo or azithromycin 500 mg 3 days a week for 6 months for adults with SCD who have FEV1<80%.

To assess acceptability of this intervention, investigators will measurement recruitment rate, retention and adherence to the study medication. Recruitment will be assessed by proportion of eligible participants that agree to be randomized. Retention will be measured as proportion randomly allocated who complete the trial. Dropout due to toxicity will be categorized using a questionnaire. Medication adherence will be assessed using the previously validated 8 item modified Morisky medication adherence scale (MMAS-8), where responses are categorized: high adherence (8 points), average adherence (6-7 points), and poor adherence (0-5 points). If recruitment rate is < 60%, the retention rate < 80%, or average adherence rate is ≤5 points, the original protocol will be examined and alternative strategies to enhance recruitment, retention, and adherence will be considered.

Specific aim 2: To evaluate the effect of 6 months of low dose azithromycin therapy on FEV1 and respiratory symptoms in patients with SCA. Baseline FEV1 testing with a portable, in-office spirometer will be completed at study enrollment and at the end of the study period (6 months). The previously validated American Thoracic Society (ATS-DLD-78 for adults) questionnaire will also be used to evaluate respiratory symptoms at baseline and end of the study. Under a separate protocol, investigators will calculate the coefficient of variation for FEV1% predicted in adults with sickle cell disease in order to define the within-subject variability for tests of respiratory function in this specific population, which has not been previously described within the medical literature. Calculation of the coefficient of variation for FEV1 % predicted will be essential for the interpretation of clinically and statistically meaningful changes in spirometry for participants who are treated with azithromycin to improve their baseline pulmonary function when compared to controls.

ELIGIBILITY:
Inclusion criteria:

1. Established diagnosis of sickle cell disease (HbSS, HbSC, HbS/β+, HbS/β0)
2. Age between 18-50 years
3. FEV1 < 80% predicted
4. Willingness to make return visits and availability by telephone for the duration of the study.

Exclusion criteria:

1. Acute respiratory symptoms
2. FEV1>80%
3. Inability to swallow pills
4. Hypersensitivity to macrolides.
5. History of cardiac arrhythmias
6. Prolonged QTc interval (>500 ms) at on baseline EKG
7. Baseline impairment of hearing by pure tone audiometry defined as patients with age-adjusted hearing thresholds >95th percentile at any one frequency of 500, 1000, 2000 and 4000 Hz.
8. The presence of a diagnosis other than SCD that results in the patient being medically unstable, or having a predicted life expectancy less than 1 year.
9. Special patient groups: prisoners, pregnant women, institutionalized patients
10. Women who are at risk of becoming pregnant during the study, and who refuse to use an acceptable means of birth control (hormonal based oral, intrauterine device or barrier contraception) for the duration of the study.
11. Patients taking tacrolimus, pimozide, disopyramide, cyclosporine, nelfinavir, bromocriptine, or hexobarbital.
12. Patients taking any medications that prolong QTc interval.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the trial will be assessed by the modified Morisky Medication Adherence Scale (MMAS - 8) | 6 months
  Acceptability of the trial will be measured based on three outcomes: recruitment, retention, and adherence rates to therapy. Retention defined as the number of participants that complete the entire study. Recruitment defined as the number of eligible participants that elect to consent to continue with study evaluations. Adherence rate measured based on MMAS score, which was previously validated in children with sickle cell disease (SCD) and scored as follows: high adherence (8 points), average adherence (6 to 7 points) and poor adherence (0 - 5 points).

SECONDARY OUTCOMES:
Change in FEV1 % predicted in response to 6 months of low dose azithromycin therapy | 6 months
Change in respiratory symptom score (by ATS-DLD-78) in response to 6 months of low dose azithromycin therapy | 6 months
Change in quality of life (by SF-36) in response to 6 months of low dose azithromycin therapy | 6 months
Number of participants with treatment-related adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. DeBaun, M.D., M.P.H., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Platt OS, Brambilla DJ, Rosse WF, Milner PF, Castro O, Steinberg MH, Klug PP. Mortality in sickle cell disease. Life expectancy and risk factors for early death. N Engl J Med. 1994 Jun 9;330(23):1639-44. doi: 10.1056/NEJM199406093302303. PMID 7993409
- [Background] Bunn HF. Pathogenesis and treatment of sickle cell disease. N Engl J Med. 1997 Sep 11;337(11):762-9. doi: 10.1056/NEJM199709113371107. No abstract available. PMID 9287233
- [Background] Vichinsky EP, Neumayr LD, Earles AN, Williams R, Lennette ET, Dean D, Nickerson B, Orringer E, McKie V, Bellevue R, Daeschner C, Manci EA. Causes and outcomes of the acute chest syndrome in sickle cell disease. National Acute Chest Syndrome Study Group. N Engl J Med. 2000 Jun 22;342(25):1855-65. doi: 10.1056/NEJM200006223422502. PMID 10861320
- [Background] Gladwin MT, Sachdev V, Jison ML, Shizukuda Y, Plehn JF, Minter K, Brown B, Coles WA, Nichols JS, Ernst I, Hunter LA, Blackwelder WC, Schechter AN, Rodgers GP, Castro O, Ognibene FP. Pulmonary hypertension as a risk factor for death in patients with sickle cell disease. N Engl J Med. 2004 Feb 26;350(9):886-95. doi: 10.1056/NEJMoa035477. PMID 14985486
- [Background] Machado RF, Hildesheim M, Mendelsohn L, Remaley AT, Kato GJ, Gladwin MT. NT-pro brain natriuretic peptide levels and the risk of death in the cooperative study of sickle cell disease. Br J Haematol. 2011 Aug;154(4):512-20. doi: 10.1111/j.1365-2141.2011.08777.x. Epub 2011 Jun 21. PMID 21689089
- [Background] Boyd JH, Macklin EA, Strunk RC, DeBaun MR. Asthma is associated with increased mortality in individuals with sickle cell anemia. Haematologica. 2007 Aug;92(8):1115-8. doi: 10.3324/haematol.11213. PMID 17650441
- [Background] Field JJ, DeBaun MR. Asthma and sickle cell disease: two distinct diseases or part of the same process? Hematology Am Soc Hematol Educ Program. 2009:45-53. doi: 10.1182/asheducation-2009.1.45. PMID 20008181
- [Background] Kassim AA, Payne AB, Rodeghier M, Macklin EA, Strunk RC, DeBaun MR. Low forced expiratory volume is associated with earlier death in sickle cell anemia. Blood. 2015 Sep 24;126(13):1544-50. doi: 10.1182/blood-2015-05-644435. Epub 2015 Aug 10. PMID 26261241
- [Background] Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL, Culver BH, Enright PL, Hankinson JL, Ip MS, Zheng J, Stocks J; ERS Global Lung Function Initiative. Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012 Dec;40(6):1324-43. doi: 10.1183/09031936.00080312. Epub 2012 Jun 27. PMID 22743675
- [Background] Bakheit AH, Al-Hadiya BM, Abd-Elgalil AA. Azithromycin. Profiles Drug Subst Excip Relat Methodol. 2014;39:1-40. doi: 10.1016/B978-0-12-800173-8.00001-5. PMID 24794904